CLINICAL TRIAL: NCT02901886
Title: REU-stop - Effect of Intensive Smoking Cessation Intervention on Smoking Cessation and Disease Activity in Patients With Rheumatoid Arthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: The Danish Rheumatism Association (Other); The Novo Nordic Foundation (Other); Region Capital Denmark (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Bente Appel Esbensen, Senior Researcher, Associate professor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-16022001
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Smoking Cessation; Disease Activity; Clinical Prevention
MeSH Terms: conditions — Arthritis, Rheumatoid; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive smoking cessation intervention (Experimental): The intervention includes 1) Individual motivational counseling in combination with 2) nicotine replacement therapy.
  The intervention consists of five individual motivational counselling sessions, each lasting 20 to 40 minutes over a period of six weeks with a trained smoking cessation counsellor. The principles of motivational counselling are based on the trans theoretical model of change. The smoking cessation counsellor has also been trained in motivational counselling techniques specific to this intervention.
  2. Nicotine replacement therapy The participants in the intervention group will be offered nicotine replacement therapy (NRT) free of charge and if accepted it will be tailored individually according to the Fagerström's Test for Nicotine Dependence.
  The participants will note their tobacco and NRT consumption in a smoking diary.
  Interventions: Behavioral: Intensive smoking cessation intervention
- Control (No Intervention): The control group will receive the standard treatment and care in the rheumatology outpatient clinic. The participants will be encouraged to write a diary describing their tobacco use during the trial period. If participants in the control group express an interest in receiving smoking cessation counselling, they will be informed about municipal programs.

INTERVENTIONS:
Behavioral: Intensive smoking cessation intervention — The intervention includes 1) Individual motivational counseling (5 meetings within 6 weeks) in combination with 2) nicotine replacement therapy.
  Arms: Intensive smoking cessation intervention

SUMMARY:
This study aims to test the effect of an intensive smoking cessation intervention (motivational counseling combined with nicotine replacement) on smoking cessation and disease activity in patients with Rheumatoid Arthritis (RA). Half of the patients will participate in a smoking cessation intervention; the other half will receive usual treatment.

DETAILED DESCRIPTION:
Tobacco smoking is a well-known environmental risk factor for developing rheumatoid arthritis (RA). The onset of RA can occur in all age groups, with the majority being women aged 50-60 years. RA is a chronic inflammatory disease and cannot be cured. However, the activity of the disease can be reduced by medication. During periods with high disease activity, patients experience increased pain and fatigue and subsequent restrictions in social life, psychical activity and activities of daily life. Furthermore, the inflammatory process underlying RA can cause pain, fatigue, reduced health-related quality of life and reduced physical function. Patients with RA are at increased risk of cardiovascular diseases similar to the risk demonstrated in patients with diabetes. Furthermore, several studies indicate that smokers with inflammatory arthritis tend to experience more pain and fatigue, and a reduced quality of life compared to non-smokers.

Aim: This randomized controlled trial (RCT) in patients with RA aims to examine the effect of intensive smoking cessation intervention (motivational counselling combined with tailored nicotine replacement therapy) versus standard care on smoking cessation, and consequently on disease activity. Secondary objectives are to explore the effect on flare, risk factors for CVD, lung function, physical function, HR-QoL, pain and fatigue in patients with RA.

Material and Methods Trial design: The trial is an international, multicentre, randomized RCT in which daily smokers with RA in remission or with low-moderate disease activity ≤ 5.1 DAS28 (Disease Activity Score - based on 28 joints assessment, serum-C-reactive protein (CRP) and patient's Global assessment of a visual analogue scale (VAS)) will be randomized 1:1 to either an intervention group or to a control group. Patients will be followed for 58 weeks, including the 6-week intervention period and 3 months, 6 months and 12 months into the post-intervention follow-up period.

Study setting: We will recruit patients from the Center for Rheumatology and Spine Diseases, Rigshospitalet, Denmark and from the Preventive Cardio-Rheuma Clinic, Department of Rheumatology, Diakonhjemmet Hospital, Oslo, Norway.

Randomization and blinding: Immediately after collecting baseline data using stratified block randomization (block size 6-10) participants will be randomized to either 1) the intervention group or 2) the control group. The stratification variables are trial site and Anti-cyclic citrullinated peptide (Anti-CCP status). The allocation sequence is generated using computer-generated random numbers. Participants will be informed about their group allocation directly after randomization. For participants randomized to the smoking cessation intervention group, the first intervention meeting will be scheduled as soon as possible, preferably immediately after randomization. It is not possible either to blind participants to their allocated intervention or to blind the project nurses performing the intervention. The primary outcomes will be assessed by blinded assessors and smoking cessation will be self-reported by participants and validated biochemically.

Data collection:All outcomes are assessed at three months (18 weeks post-intervention), 6 months (30 weeks post-intervention) and 12 months follow-up (58 weeks post-intervention).

We will retrieve data from the DANBIO database regarding the participants' pharmacological treatment, duration of RA, CRP levels, IgM rheumatoid factor and Anti-CCP status. Additional descriptive data include participants' demography, socio economic situation, lifestyle (smoking and alcohol) and consumption of pain killers obtained via a questionnaire. Co-morbidities are assessed using the Charlson's Co-morbidity Scale obtained from the electronic patient journal.

All participant-reported questionnaires will be completed electronically on a tablet connected to DANBIO, which will be used only for participants in the trial. Blood samples will be destroyed immediately after the analyses are done.

All outcomes excluding patient-reported outcomes will be assessed by project nurses blinded to the patients' group allocation.

Ethics, confidentiality and dissemination: The trial will be carried out in accordance with the Helsinki Declaration. The project has been approved by The Regional Committee on Health Research Ethics (H-16022001) and the Danish Data Protection Agency (I-suite number 04849). The trial has been reported to Clinicaltrials.gov (NCT02901886). All data and information collected during the trial will be kept confidential and in accordance with the requirements of the Danish and Norwegian Data Protection Agencies and Good Clinical Practice.

ELIGIBILITY:
Inclusion criteria Patients will be included in the study if they have RA as defined by the American College of Rheumatology (ACR) 1987 criteria and/or European League Against Rheumatism (EULAR) 2010 criteria (32, 33), >18 years of age, smoking tobacco daily, are able to understand and speak Danish or Norwegian, respectively. Furthermore, patients need to for the past three months to have been in clinical remission or low-moderate disease activity (DAS28 ≤ 5.1) and in stable anti-rheumatic medical treatment as documented in 1) the DANBIO registry in Denmark, or 2) the electronic patient journal, Department of Rheumatology, Diakonhjemmet Hospital, Oslo, Norway.

Exclusion criteria Patients will be excluded from the study if they have had a change of dose or preparation in anti-rheumatic medical treatment within the previous 3 months, or a scheduled change in anti-rheumatic medical treatment, including glucocorticoid injection during the previous month, are cognitively or otherwise unable to give informed consent, are pregnant or breastfeeding.

Excluded patients, and eligible patients who do not want to participate, will be registered in one of the following three categories 1) not meeting the inclusion criteria 2) refused to participate 3) other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported continuous smoking cessation validated by exhaled carbon-monoxide at 3 months follow-up | 3 months post-intervention
  The participants' smoking status will be monitored by self-reported continuous smoking cessation validated by exhaled carbon monoxide (CO) in breath (CO-Check, NEOMED GmbH; Germany). Carbon monoxide values > 10 parts per million (ppm) indicate tobacco smoking
EULAR clinical response (an improvement in DAS28 of >0.6) at 3 months follow-up | 3 months post-intervention
  The recommended EULAR clinical response in relation to disease activity will be assessed using DAS28 at 3 months post-intervention. The DAS28 score consists of four elements; CRP, number of swollen joints, number of painful joints (maximum 28) and a Global General Health VAS score. The joint count and Global General Health are assessed by both the participant and a project nurse blinded to group allocation

SECONDARY OUTCOMES:
Self-reported smoking status at 6 and 12 months post-intervention | 6 and 12 months post-intervention
  Smoking status will be monitored by self-reported continuous smoking cessation and biochemically validated by exhaled CO. Continuous smoking cessation will be measured by asking the patients who reports 7-day point prevalence (7 day time-line follow back) how many days they have not been smoking. Smoking status information is self-reported by the participant and documented in the smoking diary at 3 months post intervention (week 18). To be grouped as having "stopped smoking" both self-reported and biochemical analysis should indicate this.
EULAR repsonse at 6 and 12 months post-intervention | 6 and 12 months post-intervention
  Disease activity will be registered by DAS28, as described above in primary outcome.
Disease activity measured by DAS28 at 3, 6 and 12 months post-intervention | 3, 6 and 12 months post-intervention
  DAS28 as described above.
Change in number of swollen and tender joints at 3, 6 and 12 months post-intervention | 3, 6 an 12 months post-intervention
  Assessed by a person blinded to the intervention
Physician and patient Global VAS | 3, 6 and 12 months post-intervention
  Assessed by a person blinded to the intervention
C-reactive protein (CRP) | 3, 6 and 12 months post-intervention
  Measured using blood sample.
Patient assessed disease activity by the FLARE Instrument | 3, 6 and 12 months post-intervention
  Participants will be asked to answer the FLARE instrument (FI), which is a patient self-assessment questionnaire for detecting changes in disease activity among patients with RA. It is designed to detect both past and present disease activity. The questionnaire consists of 12 questions answered on a Likert scale (0 = completely agree, 10 = completely disagree). Higher scores indicate flare. A score > 2.5 indicates a flare.
Blood pressure and pulse | 3, 6 and 12 months post-intervention
  • Blood pressure (mmHg) and heart rate (beats/min) will be measured after 5 minutes of rest (supine position) (Mobil-O-Graph, IEM; Germany). If it exceeds 140/90 mmHg, two additional measurements will be performed and the mean of the last two will be registered.
Arterial stiffness | 3, 6 and 12 months post-intervention
  • Arterial stiffness will be measured by pulse wave velocity (PWV) (Mobil-O-Graph, IEM; Germany). High PWV is defined as > 9.9 m/s
Serum lipids | 3, 6 and 12 months post-intervention
  Serum lipids (TC, HDL-c, LDL-c and TG) will be measured in venous blood samples.
HbA1c | 3, 6 and 12 months post-intervention
  Will be measured using blood sample.
Waist circumference | 3, 6 and 12 months post-intervention
  • Waist circumference will be evaluated by a tape measure in centimetres (cm) while the patient is standing. For women with a waist circumference >80 cm there is an increased risk of CVD while the risk is further increased for waist circumference >88 cm. For men the measures are defined as >94 cm and >102 cm, for increased, and further increased, risk of CVD, respectively.
Body weight | 3, 6 and 12 months post-intervention
  • Body weight will be measured to the nearest 0.1 kg (with ordinary clothes, but without shoes) (OBH Nordica, Slim Light, 150 kg, Taastrup Denmark).
Lung function | 3, 6 and 12 months post-intervention
  FEV1 will be measured by spirometer (EasyOneTM, Model 2001 diagnostic Spirometer, Model 2010 Cradle, NDD Medizintechnik AG; Switzerland).
Physical function | 3, 6 and 12 months post-intervention
  HAQ is a standardized questionnaire for assessing disability and physical function in patients with RA. The instrument contains 20 items with four possible answers in eight categories; dressing, rising from a seat, eating, walking, personal hygiene, stretching for an object, grabbing an object and everyday activities. The questionnaire also includes VAS scales for pain, fatigue and general health. In DANBIO five additional questions have been added. They also have four possible answers and relate to physical function, sleep, anxiety and depression. In this study we will use the 25 questions as used in DANBIO.
Health-related quality of life | 3, 6 and 12 months post-intervention
  HR-QoL is measured using the following two questionnaires:
  1. SF-36 is a generic instrument measuring HR-QoL by 36 items on eight scales. The scales are; physical function, physical activity, limitations, pain, general health, vitality, social function, emotional activity limitations and mental health; they are summarized in two summary scales; 1) the physical component scale (PCS) and 2) the mental component scale (MCS).
  2. The questionnaire contains five items (movement, personal care, usual activities, pain and anxiety/depression) each with five possible ratings.
Pain Pain | 3, 6 and 12 months post-intervention
  Pain related to RA is self-reported by participants using the VAS. Participants rate their subjectively experienced level of pain from 0-10. Zero represents "no pain" and 10 represent the "worst imaginable pain". The scale is included in HAQ.
Fatigue | 3, 6 and 12 months post-intervention
  The BRAF-NRS assesses fatigue in patients with RA. It includes three questions concerning fatigue (level, effect and coping) over the previous seven days. Participants rate fatigue on a scale from 0-10 . Zero represent "no fatigue" and 10 represent the "worst fatigue".

CONTACTS AND LOCATIONS:
Locations (2):
- Center for Rheumatology and Spine Diseases, Rigshospitalet, Glostrup Municipality, Denmark
- Preventive Cardio-Reuma Clinic, Diakonhjemmet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Esbensen BA, Thomsen T, Roelsgaard IK, Ostergaard M, Hetland ML, Andersen L, Tonnesen H, Semb AG, Christensen R. Effect of an intensive smoking cessation intervention on smoking cessation and disease activity in patients with rheumatoid arthritis: a randomised controlled trial. Rheumatology (Oxford). 2025 Aug 21:keaf448. doi: 10.1093/rheumatology/keaf448. Online ahead of print. PMID 40839209
- [Derived] Roelsgaard IK, Thomsen T, Ostergaard M, Christensen R, Hetland ML, Jacobsen S, Andersen L, Tonnesen H, Rollefstad S, Semb AG, Esbensen BA. The effect of an intensive smoking cessation intervention on disease activity in patients with rheumatoid arthritis: study protocol for a randomised controlled trial. Trials. 2017 Nov 28;18(1):570. doi: 10.1186/s13063-017-2309-5. PMID 29183347